CLINICAL TRIAL: NCT00981994
Title: Development, Implementation, and Evaluation of Novel Strategies to Reduce Inappropriate Antimicrobial Use in Community and Healthcare Settings
Brief Title: Evaluation of an Algorithm to Reduce Antibiotic Prescribing for Acute Bronchitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: University of California, San Francisco (Other); Geisinger Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5R01CI000611 (NIH)
Record Dates: First submitted 2009-09-14; First posted 2009-09-22 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-11

CONDITIONS: Acute Respiratory Tract Infection
Keywords: respiratory infection; antimicrobial drugs; decision support; Adult patients
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Electronic Decision Support (Experimental): Use of electronic decision support to provide the treatment algorithm for providers managing patients with acute respiratory infections.
  Interventions: Behavioral: Decision Support for ARI Management
- Paper Decision Support (Experimental): Use of paper based tools to provide the treatment algorithm for providers managing patients with acute respiratory infections.
  Interventions: Behavioral: Decision Support for ARI Management
- Usual Care (No Intervention): Usual Care

INTERVENTIONS:
Behavioral: Decision Support for ARI Management — Use of history and physical examination findings to estimate probability of pneumonia in patients with acute respiratory infections and thereby guide treatment decisions
  Arms: Electronic Decision Support; Paper Decision Support

SUMMARY:
Inappropriate use of antibiotics to treat patients with acute bronchitis is a significant factor contributing to the selection of antimicrobial drug resistant pathogens, which threaten the effectiveness of available therapies to treat common community-acquired bacterial infections. A key factor driving overuse of antibiotics is inaccurate estimation of pneumonia risk among patients with acute cough illnesses. This study will use a cluster randomized trial design within the Geisinger Health System's integrated clinic network to measure the efficacy of an algorithm driven clinical decision support tool to safely reduce the frequency of unnecessary antibiotic prescriptions for adult patients with lower respiratory tract infections.

DETAILED DESCRIPTION:
The rapid rise in antibiotic resistance among common bacteria are adversely affecting the clinical course and health care costs of community-acquired infections. Because antibiotic resistance patterns are strongly correlated with antibiotic use patterns, multiple organizations have declared reductions in unnecessary antibiotic use to be critical components of efforts to combat antibiotic resistance. Among humans, the vast majority of unnecessary antibiotic prescriptions are used to treat acute respiratory tract infections (ARIs) that have a viral etiology. In particular, despite the fact that numerous controlled trials have demonstrated no benefit of antibiotic therapy for patients with acute bronchitis, the majority of patients diagnosed with acute bronchitis continue to receive antibiotic therapy across diverse treatment settings. Recently, the National Committee on Quality Assurance adopted the proportion of adult visits diagnosed as acute bronchitis when an antibiotic was NOT prescribed as a quality measure within the HEDIS data set. Recent results from the HEDIS dataset emphasize the continued high rates of antibiotic prescribing for patients with acute bronchitis. One key factor driving overuse of antibiotics in the management of patients with lower respiratory tract infections-such as acute bronchitis-is diagnostic uncertainty and inaccurate risk estimation of underlying pneumonia in such patients. Recently, our study team has observed substantial reductions in antibiotic prescribing following the incorporation of a diagnostic and treatment algorithm into an acute care setting. This acute cough management algorithm incorporates data on vital signs and symptoms distinguishing patients with community-acquired pneumonia from other patients with acute cough illness, specifically those with acute bronchitis. The acute cough management algorithm has become even more valuable in recent years due to the introduction of quality measures that emphasize the timely administration of antibiotics for patients with community-acquired pneumonia. Thus, strong empirical evidence of the effectiveness of such an algorithm could lead to wide adoption of the algorithm and substantial improvements in antibiotic prescribing. The investigative team is proposing a unique partnership with Geisinger Health System, a large integrated health network, to implement and evaluate the algorithm. Utilizing a cluster-randomized trial design across 33 practice sites, we will address the following aims: 1) To measure the reduction in antibiotic prescribing resulting from incorporation of the algorithm compared to usual care sites utilizing two different implementation strategies, one poster-based and one electronic health record-based, 2) To measure revisits, delayed hospitalizations and net economic costs associated with algorithm implementation, and 3) To evaluate local practice characteristics influencing the level of implementation and ultimate performance success at intervention sites. In a final component of the study, the investigators will partner with NCQA to disseminate study results through the national network of participating plans and stimulate wide spread adoption of the algorithm and quality improvement methods.

ELIGIBILITY:
Inclusion Criteria:

* Primary care practice sites within the Geisinger Health System

Exclusion Criteria:

* Sites with < 1000 visits per year for acute respiratory infection

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3300 (Actual)
Dates: Start 2009-10; Primary Completion 2011-05 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Proportion of visits to primary care clinic associated with antibiotic prescriptions | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Joshua P Metlay, MD, PhD, Principal Investigator — University of Pennsylvania; Ralph Gonzales, MD,MS, Principal Investigator — University of California, San Francisco

REFERENCES:
- [Derived] Gonzales R, Anderer T, McCulloch CE, Maselli JH, Bloom FJ Jr, Graf TR, Stahl M, Yefko M, Molecavage J, Metlay JP. A cluster randomized trial of decision support strategies for reducing antibiotic use in acute bronchitis. JAMA Intern Med. 2013 Feb 25;173(4):267-73. doi: 10.1001/jamainternmed.2013.1589. PMID 23319069